CLINICAL TRIAL: NCT00729430
Title: Prognostic, Anti-arrhythmic, and Ventricular Remodeling Effects of High Dose Fish Oil in Patients With a Recent Myocardial Infarction
Brief Title: Effect of High Dose Fish Oil Supplementation After Recent Heart Attack Using Magnetic Resonance Imaging
Acronym: OmegaREMODEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Raymond Y. Kwong, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 591; R01HL091157-01 (NIH)
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Myocardial Infarction; Death, Sudden, Cardiac
Keywords: Heart Attack; Sudden Cardiac Death; Peri-infarct Zone; Omega-3 Fatty Acids; Biological Markers; Cytogenetic Analysis; Cardiac Arrest
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden, Cardiac; Heart Arrest | interventions — Fatty Acids, Omega-3; Omacor; halofantrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 Fatty Acids (Experimental): Participants will receive a highly purified form of omega-3 fatty acids for 6 months.
  Interventions: Drug: Omega-3 Fatty Acids (Fish Oil Supplements)
- Placebo (Placebo Comparator): Participants will receive placebo for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 Fatty Acids (Fish Oil Supplements) — 4 grams of omega-3 fatty acids taken orally once per day for 6 months
  Other Names: Lovaza (GlaxoSmithKline)
  Arms: Omega-3 Fatty Acids
Drug: Placebo — Placebo tablets taken orally once per day for 6 months
  Other Names: Corn oil placebo
  Arms: Placebo

SUMMARY:
Doctors use magnetic resonance imaging (MRI) to obtain detailed pictures of the inside of the body. This study will evaluate a new MRI technique in people who have recently had a heart attack. Researchers will also examine the effect of fish oil supplementation on heart health in study participants.

DETAILED DESCRIPTION:
A new MRI technique to examine the heart was recently developed. In this study, researchers will use this new technique to evaluate the heart in people who have recently had a heart attack to determine whether a specific pattern of heart muscle damage is related to sudden cardiac death. This fatal condition, also known as cardiac arrest, occurs when the heart abruptly stops pumping blood to the body, resulting in loss of consciousness, absence of pulse, and a stop in breathing. The most common cause of sudden cardiac death is a heart attack.

In addition to evaluating the new heart MRI technique, this study will also examine the effects of fish oil supplementation in people who have recently had a heart attack. Recent research has shown that omega-3 fatty acids, commonly found in fish oil, may be beneficial for people with heart conditions. Lastly, the study will determine whether specific biomarkers and genetic factors can help predict the likelihood of a person dying from sudden cardiac death after previously experiencing a heart attack.

Apart from studying the likelihood of sudden cardiac death, This study will measure the change in structure and pumping function of the heart (known as ventricular remodeling) and this study will determine if the high dose of fish oil treatment will result in an improvement of the heart.

This study will enroll people who have had a heart attack in the 2 to 4 weeks before study entry. At a baseline study visit, participants will undergo an MRI of their heart and complete an exercise stress test on a treadmill. A blood sample will be collected, and women will provide a urine sample for a pregnancy test. Questionnaires asking about diet, medical history, and emotions will also be completed. Participants will then be randomly assigned to receive either fish oil supplements or placebo on a daily basis for 6 months. Every 2 to 3 months, study researchers will call participants to check on their health and progress. At a study visit at Month 6, participants will undergo repeat baseline testing. After this visit, study researchers will call participants every 6 months for 3 years to follow up on participants' health status.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a heart attack in the 2 to 4 weeks before study entry
* Lives in the greater Boston area or adjacent regions (within a 50-mile radius of Boston)

Exclusion Criteria:

* Unable to undergo an MRI because of metallic implants (e.g., pacemakers, an implantable cardioverter defibrillator [AICD]) at time of study entry
* Active cancer or any other terminal illness with an expected survival rate of less than 6 months after study entry
* Significant kidney dysfunction with a glomerular filtration rate (GFR) of less than 60 mL/min in the 2 weeks before study entry
* Inability to follow study procedures
* Pregnant
* Hemodynamic instability
* Urgent clinical need for a pacemaker or AICD
* Inaccessibility of medical records

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2008-08; Primary Completion 2013-10 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Y. Kwong, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Shapiro Cardiovascular Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data with GISSI Heart Failure group for pooling and meta-analysis

REFERENCES:
- [Background] Yan AT, Shayne AJ, Brown KA, Gupta SN, Chan CW, Luu TM, Di Carli MF, Reynolds HG, Stevenson WG, Kwong RY. Characterization of the peri-infarct zone by contrast-enhanced cardiac magnetic resonance imaging is a powerful predictor of post-myocardial infarction mortality. Circulation. 2006 Jul 4;114(1):32-9. doi: 10.1161/CIRCULATIONAHA.106.613414. Epub 2006 Jun 26. PMID 16801462
- [Result] Heydari B, Abdullah S, Pottala JV, Shah R, Abbasi S, Mandry D, Francis SA, Lumish H, Ghoshhajra BB, Hoffmann U, Appelbaum E, Feng JH, Blankstein R, Steigner M, McConnell JP, Harris W, Antman EM, Jerosch-Herold M, Kwong RY. Effect of Omega-3 Acid Ethyl Esters on Left Ventricular Remodeling After Acute Myocardial Infarction: The OMEGA-REMODEL Randomized Clinical Trial. Circulation. 2016 Aug 2;134(5):378-91. doi: 10.1161/CIRCULATIONAHA.115.019949. PMID 27482002
- [Derived] Fujikura K, Heydari B, Ge Y, Kaneko K, Abdullah S, Harris WS, Jerosch-Herold M, Kwong RY. Insulin Resistance Modifies the Effects of Omega-3 Acid Ethyl Esters on Left Ventricular Remodeling After Acute Myocardial Infarction (from the OMEGA-REMODEL Randomized Clinical Trial). Am J Cardiol. 2020 Mar 1;125(5):678-684. doi: 10.1016/j.amjcard.2019.11.032. Epub 2019 Dec 9. PMID 31948661
- [Derived] Kwong RY, Heydari B, Ge Y, Abdullah S, Fujikura K, Kaneko K, Harris WS, Jerosch-Herold M, Antman EM, Seidman JG, Pfeffer MA. Genetic profiling of fatty acid desaturase polymorphisms identifies patients who may benefit from high-dose omega-3 fatty acids in cardiac remodeling after acute myocardial infarction-Post-hoc analysis from the OMEGA-REMODEL randomized controlled trial. PLoS One. 2019 Sep 18;14(9):e0222061. doi: 10.1371/journal.pone.0222061. eCollection 2019. PMID 31532795

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Omega-3 Fatty Acid Arm: Participants will receive a highly purified form of omega-3 fatty acids for 6 months.
  Omega-3 Fatty Acids (Fish Oil Supplements): 4 grams of omega-3 fatty acids taken orally once per day for 6 months
- Placebo Arm: Participants will receive placebo for 6 months.
  Placebo: Placebo tablets taken orally once per day for 6 months
Period: Overall Study
Arm/Group | High Dose Omega-3 Fatty Acid Arm | Placebo Arm
Started | 180 | 178
Completed | 133 | 128
Not Completed | 47 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Omega-3 Fatty Acid Arm | Placebo Arm | Total
Number analyzed (Participants) | 180 | 178 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10) | 58 (10) | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 38 | 70
  Male | 148 | 140 | 288
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 180 | 178 | 358

OUTCOME MEASURES:

1. Primary Outcome: Effect of Omega-3 Fatty Acids on Adverse Left Ventricular Remodeling
Description: Measured as change in left ventricular end-systolic volume indexed to body surface area from baseline to post-treatment (6-months)
Time Frame: Before and after study treatments
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | High Dose Omega-3 Fatty Acid Arm | Placebo Arm
Number analyzed (Participants) | 180 | 178
Percent Change | -5.4 (16.6) | 1.2 (20.9)

2. Secondary Outcome: Effect of Omega-3 Fatty Acids on Non-Infarct Myocardial Fibrosis
Description: Measured as change in myocardial extracellular volume fraction of non-infarcted myocardium from baseline to post-treatment (6-months)
Time Frame: Measured in the 3-year follow-up period after participant's last study visit
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | High Dose Omega-3 Fatty Acid Arm | Placebo Arm
Number analyzed (Participants) | 180 | 178
Percent Change | -2.1 (14) | 3.4 (15)

3. Secondary Outcome: Effect of Omega-3 Fatty Acids on Left Ventricular Ejection Fraction
Description: Measured as change in left ventricular ejection fraction from baseline to post-treatment (6-months)
Time Frame: Measured in the 3-year follow-up period after participant's last study visit
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- High Dose Omega-3 Fatty Acids Arm: Participants will receive a highly purified form of omega-3 fatty acids for 6 months.
  Omega-3 Fatty Acids (Fish Oil Supplements): 4 grams of omega-3 fatty acids taken orally once per day for 6 months
Arm/Group | High Dose Omega-3 Fatty Acids Arm | Placebo Arm
Number analyzed (Participants) | 180 | 178
Percent Change | 4.8 (11) | 2.1 (12)

4. Secondary Outcome: Effect of Omega-3 Fatty Acids on Infarct Size
Description: Measured as change in infarct size from baseline to post-treatment (6-months)
Time Frame: Measured in the 3-year follow-up period after participant's last study visit
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | High Dose Omega-3 Fatty Acids Arm | Placebo Arm
Number analyzed (Participants) | 180 | 178
Percent Change | -8.8 (39.9) | -1.9 (57.7)

ADVERSE EVENTS:
Time Frame: Measured in the 3-year follow-up period after participant's last study visit
Description: Adverse events were evaluated every 2 months during the 6-month study drug period by an investigator with conducted scripted telephone interviews with each patient. Tolerance to study drug, adverse events, and pill counts were also evacuated during these interviews.
Arm/Group | High Dose Omega-3 Fatty Acids Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 1/180 | 0/178
Other Adverse Events (participants affected / at risk) | 18/180 | 11/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Omega-3 Fatty Acids Arm (N=180) | Placebo Arm (N=178)
Allergic Reaction (Tongue Swelling) (Immune system disorders) | 1 (1) | 0 (0) — One omega-3 fatty acid treated patient experienced tongue swelling 1 month after enrollment that necessitated study drug termination, which resulted in resolution of the patient's symptoms.
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) — Clinically significant bleeding or drop in hematocrit levels.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Omega-3 Fatty Acids Arm (N=180) | Placebo Arm (N=178)
Fishy Taste in Mouth (Gastrointestinal disorders) | 8 (8) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (10) | 9 (9)

LIMITATIONS AND CAVEATS:
The study was not powered to evaluate for clinical heart failure and hard cardiac outcomes. A prospective trial would be necessary to determine the effect of earlier and high-dose omega-3 fatty acid therapy on improving clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No